CLINICAL TRIAL: NCT04812847
Title: Infecciones Por patógenos Gramnegativos Con Multirresistencia a Drogas en Neonatos de Alto Riesgo en el Noreste de México
Brief Title: Multidrug Resistant Gram-negative Pathogen Infections in High Risk Neonates in the Northeast of Mexico
Acronym: InfGNMDR-Neo
Status: Completed | Type: Observational
Sponsor: Instituto Tecnologico y de Estudios Superiores de Monterey (Other)
Responsible Party: Principal Investigator, Victor Javier Lara-Diaz, M.D., Ph.D., Professor-Researcher, Instituto Tecnologico y de Estudios Superiores de Monterey
Other Study IDs: InfGNMDR-Neo
Record Dates: First submitted 2021-03-10; First posted 2021-03-24 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Infant Newborn Disease
Keywords: Drug Resistance, Multiple, Bacterial.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Isolated microorganism, recovered from culture plates, cryo-preserved at -80°C media until analysis, and thawed and seeded onto EMB (Eosin-Methylene Blue) agar plates, will be used for qrtPCR (quantitative real-time Polimerase Chain reaction)amplification of fragments of genes of interest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gram negative infection, MDR present: Neonates with one or more gram-negative bacterial isolates with MDR characteristics during their clinical course in the Neonatal Intensive Care Unit of the study hospital.
  Interventions: Diagnostic Test: Identification of MDR characteristics
- Gram negative infection, MDR absent: Neonates with one or more gram-negative bacterial isolates with no MDR characteristics during their clinical course in the Neonatal Intensive Care Unit of the study hospital.
  Interventions: Diagnostic Test: Identification of MDR characteristics

INTERVENTIONS:
Diagnostic Test: Identification of MDR characteristics — Identification of MDR in culture media, followed by amplification of related genes from the bacterial isolates

SUMMARY:
The main objective of this project is to establish a prospective cohort to measure the Gram-negative infection burden in neonates under special care in a regional referral hospital, and to characterize all microorganisms isolates from these subjects at the phenotype and genotype level, specifically in relation to the expression of multi-drug resistance (MDR) associated genes (Molecular characterization of Gram-negative MDR isolates).

DETAILED DESCRIPTION:
The investigators propose a mixed design approach, a cohort´s study with a nested case-control analysis. Study subjects will be the gram-negative isolates at the study hospital clinical laboratory. The cohort´s exposure factor will be the presence or absence of a multidrug resistance gram-negative bacterial isolate.

The prospective cohort will allow the estimation of Gram-negative infection burden in the study population, and the characterization of all microorganisms isolates from study subjects at the phenotype and genotype level, specifically in relation to the expression of multi-drug resistance (MDR) associated genes (Molecular characterization of Gram-negative MDR isolates); the cohort will be formed by each neonate, from the admission to special care, the isolation date and then follow-up until the resolution, being it discharge either alive, dead or by transfer to another facility. Risk ratios for each of these outcomes will be calculated.

Cases-controls analysis will allow the research team to identify main risk factors present in those individuals who further had or did not have a gram-negative MDR isolate, by calculation of associated odds ratios for concurrent perinatal factors. Another project goal, to establish correlations and measure risk factors (Odds ratios) between Gram-negative infection with MDR organisms and concurrent illness and treatments offered in the special care nursery (medical [antibiotics, non-steroid anti-inflammatory drugs, steroids, others], surgical, and clinical procedures) in neonates under special care, will also be attained through the nested cases and controls study approach.

Finally, a derivative from this project will be the establishment of the North-East Mexico Regional Repository of bacterial isolates in Neonates under special care. At the first stage, this repository will preserve specimens of bacteria, both Gram-negative and Gram-positive, along with a specially developed anonymous database of the individuals hosting those infections. In the near future, the focus of this repository may expand to fungus, parasites and perhaps viral isolates preservation.

The research team has also proposed an exploratory objective, subject to budget availability, and that is the characterization and comparison of the immuno-phenotype of those individuals affected of Gram-negative infection with MDR resistant organisms, those with infection with other organisms and those not affected by infectious complications.

All gram-negative isolates will be probed for the gene expression of 38 selected antibiotic resistance loci, and 96 selected samples will be further studied by next generation sequentiation.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates of either sex, and any gestational age, admitted to the special care nursery of Hospital Regional Materno Infantil (Includes also out-born and transferred babies),
2. Treating physician´s order to draw any biological sample and send it for culture at the hospital´s clinical laboratory.
3. A culture with an isolate of Gram-negative bacteria.

Exclusion Criteria:

1. Any culture negative for bacterial growth
2. Any culture with Gram-positive bacteria, or fungus growth.

Ages: 1 Day to 180 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates, both at term and preterm, of any gestational age, under special care in the Neonatology Division of a tertiary care regional perinatal center in the Northeast of Mexico.
Sampling Method: Non-Probability Sample
Enrollment: 597 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Burden of Gram Negative organisms infections | Through study completion, an average of three months
  The isolation of a gram-negative organism, from any clinical site, in neonates under clinical care in special care nursery; Incidence = New cases during the study period, Prevalence = Total cases during the study period.

SECONDARY OUTCOMES:
Odds ratio for the occurrence of Gram-negative MDR infections | Through study completion, an average of three months
  To identify and measure the Odds-ratio for the occurrence of Gram-negative infection with MDR resistant organisms and all concurrent perinatal factors. This will be done through a nested case and controls study approach.
Risk factors for the occurrence of Gram-negative MDR infections. | Through study completion, an average of three months
  To establish correlations and measure risk factors (Relative risks) between Gram-negative infection with MDR organisms and concurrent illness and treatments offered in the special care nursery (medical [antibiotics, non-steroid anti-inflammatory drugs, steroids, others], surgical, and clinical procedures) in neonates under special care. This will be attained with a cohorts study approach.

CONTACTS AND LOCATIONS:
Overall Officials: Victor Javier Lara-Diaz, MD, PhD, Study Chair — Tecnológico de Monterrey, Escuela de Medicina y Ciencias de la Salud; Cuauhtémoc Licona-Cassani, PhD, Principal Investigator — Tecnológico de Monterrey, Centro de Biotecnología FEMSA; Marion Genevieve Brunck, PhD, Principal Investigator — Tecnológico de Monterrey, Escuela de Ingeniería y Ciencias, GIEE on Translational Omics
Locations (1):
- Hospital Regional Materno Infantil de Alta Especialidad, Secretaría de Salud, Guadalupe, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Initially, we plan to share raw data with qualified researchers and entities worldwide, but we have not yet decided a specific repository.